CLINICAL TRIAL: NCT02781779
Title: Comparison of Outcomes Between the Use of Silverlon® Dressing and AQUACEL® AG Dressing Post Cardiac Device Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas City Heart Rhythm Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003363
Record Dates: First submitted 2016-05-20; First posted 2016-05-24 (Estimated); Results first posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2020-04

CONDITIONS: Infections; Wounds and Injuries
Keywords: Cardiac Implantable Electronic Device; Implant
MeSH Terms: conditions — Infections; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Silverlon® (Active Comparator): Subjects randomized to this arm will receive Silverlon® dressing postoperative.
  Interventions: Device: Silverlon®
- AQUACEL® AG (Active Comparator): Subjects randomized to this arm will receive AQUACEL® AG dressing postoperative.
  Interventions: Device: AQUACEL® AG

INTERVENTIONS:
Device: Silverlon® — Silverlon wound dressings
  Arms: Silverlon®
Device: AQUACEL® AG — AQUACEL® AG wound dressings
  Arms: AQUACEL® AG

SUMMARY:
The purpose of this study is to learn how effective each of the two dressings, Silverlon® and AQUACEL® AG, are in preventing post cardiac implantable electronic devices (CIED) procedure wound infections.

DETAILED DESCRIPTION:
This is a single center, prospective, 2-arm randomized, non-blinded study. A total of 100 participants will be assigned to the Silverlon arm and 100 to the AQUACEL AG arm.

The number of procedures to implant CIED has risen in recent years. With this rise has also brought a rise in post-procedure infections. Infections will happen and there is a continued need to improve all aspects of the surgery and post-operative care. Wound coverage with appropriate dressings is one aspect that needs to be studied in CIED implant patients. Silverlon and AQUACEL AG are two options of dressings available for these patients. This study will look to see if one of the two is a better option for post-operative CIED implant patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for a CIED implant, generator change, or upgrade at the University of Kansas Hospital
* Able to give informed consent

Exclusion Criteria:

* Patients who are already on antibiotics for another reasons
* Immunocompromised patients such as those on immunosuppressant's and HIV positive patients
* Patients who are post device explant for lead infection
* Patients with an allergy to adhesive, silver or an allergy to the dressing(s) or their components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospectively enrolled patients undergoing CIED implantation, upgrade, or generator change from June 2016-June 2017 were randomized to receive one of the two dressings at the end of the procedure.
Pre-assignment Details: Immunocompromised patients and those on non-standard antibiotic regimens were excluded.
Period: Overall Study
Arm/Group | Silverlon® | AQUACEL® AG
Started | 78 | 69
Completed | 78 | 69
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Silverlon® | AQUACEL® AG | Total
Number analyzed (Participants) | 78 | 69 | 147
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.4 (13.7) | 68.5 (14.2) | 69 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 54 | 47 | 101
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 76 | 68 | 144
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 78 | 69 | 147
body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.7 (6.3) | 29.9 (5.7) | 29.79 (6.06)
Diabetes [Count of Participants; unit: Participants] | 27 | 22 | 49
Chronic Kidney Disease (CKD) [Count of Participants; unit: Participants] | 20 | 15 | 35
Oral Anticoagulant (OAC) [Count of Participants; unit: Participants] | 33 | 32 | 65
Platelets [Mean (Standard Deviation); unit: Platelets*1000] | 210 (72) | 213 (65) | 211.41 (68.59)
Serum Creatinine (Serum Cr) [Mean (Standard Deviation); unit: mg/dL] | 1.15 (0.46) | 1.17 (0.45) | 1.16 (0.45)
International Normalized Ratio (INR) [Mean (Standard Deviation); unit: Ratio] — The INR is derived from prothrombin time (PT) which is calculated as a ratio of the patient's PT to a control PT standardized for the potency of the thromboplastin reagent developed by the World Health Organization (WHO) using the following formula:
  INR = Patient PT ÷ Control PT
  Ratio | 2 (1) | 2 (1) | 2 (0.997)

OUTCOME MEASURES:

1. Primary Outcome: Pocket Hematoma, Moderate-Severe
Description: A pocket hematoma is an accumulation of blood in or near the surgical incision which occurs because of a defect in hemostasis such as injury to blood vessels. Pocket hematoma is associated with local discomfort, an increased risk of infection, and may require surgical intervention or lead to lengthier hospital stays.
  Mild - Ecchymosis or mild effusion in the pocket, no swelling or pain to device-pocket (watchful waiting) Moderate - Large effusion in the pocket leading to swelling and causing functional impairment or pain to device-pocket Severe - Any pocket hematoma requiring: Reoperation and/or resulting in prolongation of hospitalization (defined as extended hospitalization or rehospitalization for >24 hours, postindex surgery, primarily due to hematoma) and/or requiring interruption of OAC (defined as reversal or intentional withholding, in response to pocket hematoma, resulting in subtherapeutic anticoagulation for >24 hours)
Time Frame: 7-10 days post implant
Measure: Number; unit: participants
Arm/Group | Silverlon® | AQUACEL® AG
Number analyzed (Participants) | 78 | 69
participants | 2 | 2

2. Secondary Outcome: Wound Drainage
Description: Number of participants with wound drainage
Time Frame: At time of dressing removal, up to 10 days post operative
Measure: Count of Participants; unit: Participants
Arm/Group | Silverlon® | AQUACEL® AG
Number analyzed (Participants) | 78 | 69
Participants | 1 | 1

3. Secondary Outcome: Pocket Dehiscence
Description: Pocket (Wound) Dehiscence:
  Dehiscence is a partial or total separation of previously approximated wound edges, due to a failure of proper wound healing. It may be just the surface layer or the whole wound.This scenario typically occurs 5 to 8 days following surgery when healing is still in the early stages.
Time Frame: At time of dressing removal, up to 10 days post operative
Measure: Count of Participants; unit: Participants
Arm/Group | Silverlon® | AQUACEL® AG
Number analyzed (Participants) | 78 | 69
Participants | 1 | 0

4. Secondary Outcome: Rash After Removal
Description: Number of participants with rash after dressing removal
Time Frame: At time of dressing removal, up to 10 days post operative
Measure: Count of Participants; unit: Participants
Arm/Group | Silverlon® | AQUACEL® AG
Number analyzed (Participants) | 78 | 69
Participants | 0 | 2

5. Secondary Outcome: Site Itching/Burning
Description: Number of participants with Site itching/burning
Time Frame: At time of dressing removal, up to 10 days post operative
Measure: Count of Participants; unit: Participants
Arm/Group | Silverlon® | AQUACEL® AG
Number analyzed (Participants) | 78 | 69
Participants | 7 | 4

6. Secondary Outcome: Skin Erythema
Description: Number of participants with skin erythema
Time Frame: At time of dressing removal, up to 10 days post operative
Measure: Count of Participants; unit: Participants
Arm/Group | Silverlon® | AQUACEL® AG
Number analyzed (Participants) | 78 | 69
Participants | 4 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored/assessed.
Description: Adverse events were not monitored/assessed. All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | Silverlon® | AQUACEL® AG
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT02781779/Prot_SAP_000.pdf